CLINICAL TRIAL: NCT02723747
Title: Quantitative Myocardial Perfusion Reserve by Cardiovascular Magnetic Resonance
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Ugander, MD, PhD, Karolinska Institutet
Other Study IDs: QUACK
Record Dates: First submitted 2016-03-16; First posted 2016-03-30 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Myocardial Ischemia
Keywords: myocardial ischemia; magnetic resonance imaging; perfusion; software
MeSH Terms: conditions — Myocardial Ischemia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy subjects with normal 12-lead electrocardiogram at rest.
  Interventions: Other: myocardial perfusion with magnetic resonance imaging

INTERVENTIONS:
Other: myocardial perfusion with magnetic resonance imaging

SUMMARY:
The purpose of this study is to validate a full-automated post-processing software for quantitative perfusion of the myocardium with magnetic resonance imaging.

DETAILED DESCRIPTION:
Cardiac magnetic resonance (CMR) imaging is a wide available technique for the diagnosis of myocardial ischemia. However, myocardial first-pass perfusion evaluation has been limited due to the moderate accuracy of the currently available qualitative and semiquantitative methods used to assess myocardial perfusion, and due to the lack of efficient absolute quantitative methods. Some CMR techniques and post-processing mathematical models have been developed for quantitative measurement of myocardial blood flow reserve with perfusion CMR under pharmacological stress. Measurement of these parameters with CMR have been shown to increase the accuracy of CMR in diagnosing myocardial ischemia, but most of these methods present technical challenges and have unreasonably time consuming post-processing. The aim of this study is to validate a full automated post-processing software for first pass perfusion CMR images that results in automated generated quantitative perfusion color maps.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals with normal 12-lead electrocardiogram at rest.

Exclusion Criteria:

* systolic blood pressure below 90 mmHg;
* bradycardia (< 45 heart beats/minute);
* intake of caffeine or caffeine-containing drink/medicine 24 hours prior to the examination;
* impaired renal function assessed by venous blood sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospectively enroll 80 adult healthy volunteers (40 females and 40 males).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of global myocardial first pass perfusion in mL/min/g measured in automatic post-processed color maps compared with myocardial blood volume measured in the coronary sinus (mL/min) divided by the total left ventricle mass (g) | Through study completion, an average of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ugander, MD, PhD, Principal Investigator — Department of Molecular Medicine and Surgery, Karolinska Institutet
Locations (1):
- Department of Molecular Medicine and Surgery, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nickander J, Themudo R, Thalen S, Sigfridsson A, Xue H, Kellman P, Ugander M. The relative contributions of myocardial perfusion, blood volume and extracellular volume to native T1 and native T2 at rest and during adenosine stress in normal physiology. J Cardiovasc Magn Reson. 2019 Nov 25;21(1):73. doi: 10.1186/s12968-019-0585-9. PMID 31767018